CLINICAL TRIAL: NCT06074068
Title: Examining Therapeutic Change Mechanisms in an Affect Regulation, Father-Focused Intervention for Reducing Family Violence and Associated Symptoms in Children
Brief Title: Father-Focused Intervention for Reducing Family Violence and Symptoms in Children
Acronym: F4C
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: University of Connecticut (Other); University of Delaware (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2000026789_a; 1R01HD110583-01A1 (NIH)
Record Dates: First submitted 2023-07-31; First posted 2023-10-10 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Intimate Partner Violence; Child Maltreatment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fathers for Change (Experimental): Defining features of F4C include: 1) focus on the fathering role to facilitate engagement, 2) focus on RF to understand self, partner and children and emotion regulation skills to reduce IPV and child maltreatment. F4C focuses on understanding of emotional experiences, how they impact thinking and behaviors related to partners, co-parents and children. F4C clients will meet individually with their F4C therapist for 60 minutes per week over 18 weeks.
  Interventions: Behavioral: Fathers for Change
- Duluth BIP (Active Comparator): The BIP is a psychoeducational intervention that will be delivered in 60- minute individual weekly sessions over 18 weeks. The intervention focuses on the impact of violence on victims, power and control tactics, and societal influences supporting men's violence toward women. The intervention includes didactics and experiential exercises including video vignettes and role plays to teach anger management skills.
  Interventions: Behavioral: Duluth BIP

INTERVENTIONS:
Behavioral: Fathers for Change — 18 week individual therapy focused on fathers' emotion regulation, reflective functioning and family communication.
  Arms: Fathers for Change
Behavioral: Duluth BIP — 18 week individually delivered psychoeducation and CBT focused program focused on intimate partner violence
  Arms: Duluth BIP

SUMMARY:
The goal of this clinical trial is to test the efficacy of Fathers for Change (F4C) compared to standard Batterer Intervention for fathers with a history of Intimate Partner Violence. The main question[s] it aims to answer are:

1. Is F4C more efficacious than standard BIP in reducing family violence and child mental health impairment?
2. What are the trajectories of therapeutic change targets across interventions?
3. Does father's emotion regulation and reflective functioning mediate the relationship between the two interventions and child-related outcomes? Participants will be randomized to either Fathers for Change on Batterer Intervention.

DETAILED DESCRIPTION:
Children's exposure to intimate partner violence (IPV), often perpetrated by fathers, has been described as a gateway to other adversity, with more than a 50% co-occurrence of direct forms of child maltreatment (CM). IPV exposure can wreak havoc on children, with risk for psychosocial impairments, including posttraumatic stress disorder (PTSD), that can emerge early and cascade across development. Lacking are interventions that adequately address the complex nature of IPV in families, including fatherhood and coparenting. This gap reflects a bias towards excluding offending fathers from child-focused work and an overreliance on batterer intervention programs (BIPs), which have shown negligible effects in meta-analyses and fail to address the roots of offending behaviors in fathers. Consequently, IPV exposed children remain at risk and fathers' personal and interpersonal functioning, including the father-child relationship, does not improve. In effect, there is an urgent need for effective interventions for fathers and their families. Fathers for Change (F4C) is a novel fatherhood-focused intervention with a dual focus on IPV and CM that focuses on identifying, understanding, and managing emotions to reduce aggression and improve partner and parent-child interactions. F4C has a growing evidence-base demonstrating significant reductions in family violence, improved father-child interactions, and in one open trial, improved child mental health. Proposed therapeutic mechanisms of F4C include reflective functioning (RF), the capacity for parents to understand their own and children's actions as a function of underlying states and motivations, and emotion regulation (ER), the capacity to exert control over emotional states and reactions to threat. Poor RF and ER have been associated with increased family violence and stress-related psychopathology, suggesting key focal points for intervention. To date, there have been no empirical examinations of ER and RF as therapeutic change mechanisms for reducing family violence and improving father-child interactions and child mental health. Proposed is a dual-site, multi-modal examination of ER and RF in fathers (of children 4-7 y.o.) randomized to F4C (N=180) or the Duluth Model (N=180), a BIP serving as active control. In-session observational coding will assess adaptive and maladaptive ER and RF across treatment. Weekly self-ratings will assess at-home ER and RF. Aims will (1) assess efficacy of F4C compared to a standard BIP in reducing family violence and child mental health impairment, (2) map and compare trajectories of therapeutic change targets across interventions, and (3) examine the mediating role of father's ER and RF on child-related outcomes. This proposal will grow the evidence-base for F4C and advance our understanding of therapeutic mechanisms through which F4C exerts its effects.

ELIGIBILITY:
Inclusion Criteria:

* have at least one 6 month to 12-year-old biological child with whom they have contact;
* had an incident of IPV within the last 12 months prior to screening with their child's mother (based on court/police records, coparent or self-report);
* have a currently open or recently investigated (in the last 6 months) case with CT DCF
* are able to complete assessments in English;
* agree to have their female coparents (mother of target child) contacted as collateral informants and for consent for participation of their child. If a participant has more than one child in the age range, the youngest will be selected;
* female coparents (i.e., biological mother who need not be in a relationship with the father) consents to (at minimum) provide parent-report on child; however, may opt out of child participation. If the coparent agrees to participate by providing caregiver-report on child symptoms, but declines participation of their shared child, the father may still participate in the study if he meets eligibility criteria outlined below; thus, preventing any possible retaliation against co-parents for not consenting to child participation.

Exclusion Criteria:

Fathers will be excluded based on the following exclusion criteria:

* an active full/no contact protective order pertaining to their child because this will preclude participation in the father-child play assessment (many men will have protective orders pertaining to their partners, but it is more common for men to still be allowed contact with their children);
* physiological addiction to a substance that requires detoxification. Fathers will be evaluated using the Drug Abuse Screening Test and AUDIT. If fathers report significant difficulties with physiological withdrawal (e.g., alcohol tremors or dope sickness) they will be referred for detox services. They can be re-evaluated following a detox program with documentation from the detox center of successful completion and clean urine screen;
* cognitive impairment that will not allow for understanding of the study interventions (a mini mental state score <25);
* current untreated psychotic disorder;
* currently suicidal or homicidal ideation based on screening using the BSI; or
* previously participated in F4C or a BIP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Primary participants identify as fathers. They will be targets of provided interventions. Coparents and children may be of any gender identity.
Enrollment: 1080 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Physical Intimate Partner Violence (IPV) overtime | Baseline, 19 weeks, 43 weeks and 70 weeks
  The Physical Intimate Partner Violence Subscale of the Family Socialization Interview-Revised will be used to assess physical IPV. Items are coded on a 4-point scale for severity from 0 (none) to 4 (severe). Scores are averaged to achieve a total score with a range of 0 to 4. Higher scores indicate greater frequency and severity of Physical IPV.
Change in Verbal Intimate Partner Violence (IPV) overtime | Baseline, 19 weeks, 43 weeks and 70 weeks
  The Verbal Intimate Partner Violence Subscale of the Family Socialization Interview-Revised will be used to assess verbal IPV. Items are coded on a 4-point scale for severity from 0 (none) to 4 (severe). Scores are averaged to achieve a final score with a range of 0 to 4. Higher scores indicate greater frequency and severity of verbal IPV.
Change in Physical Child Maltreatment overtime | Baseline, 19 weeks, 43 weeks and 70 weeks
  Family Socialization Interview-Revised will be used to assess physical child maltreatment. The Physical scale will be used for this outcome. Items are ranked on 0-4 point scale from 0 (none) to 4 (severe) and averaged for a final score with a range of 0 to 4 with higher scores indicating greater frequency and severity of physical child maltreatment risk.
Change in Verbal Child Maltreatment overtime | Baseline, 19 weeks, 43 weeks and 70 weeks
  Family Socialization Interview-Revised will be used to assess physical child maltreatment. The verbal scale will be used for this outcome. Items are ranked on 0-4 point scale from 0 (none) to 4 (severe) and averaged for a final score with a range of 0 to 4 with higher scores indicating greater frequency and severity of verbal child maltreatment risk.

SECONDARY OUTCOMES:
Change in Child Posttraumatic Stress Symptoms overtime | Baseline, 19 weeks, 43 weeks and 70 weeks
  The Child Trauma Symptom Checklist will be used to assess child PTSD symptoms. Each symptom item is rated according to its frequency of occurrence using a four point scale ranging from 0 ("never") to 3 ("often"). The PTSD total raw score is converted to a t-score based on measure norms with scores ranging from 0 to 100. Higher scores indicate greater severity of posttraumatic symptoms.
Change in Father-child interactions overtime | Baseline, 19 weeks, and 70 weeks
  Child interactive behavior coding based on 15 minute play assessment coded for dyadic reciprocity, fluency, conflict and hostility. Scores are on a 1 to 4 point scale. An average score is generated for a range of 1 to 4. Higher scores indicate more of the coded behavior.
Change in Coercive Controlling Intimate Partner Violence (IPV) overtime | Baseline, 19 weeks, 43 weeks and 70 weeks
  The Coercive Controlling Intimate Partner Violence Subscale of the Family Socialization Interview-Revised will be used to assess verbal IPV. Items are coded on a 4-point scale for severity from 0 (none) to 4 (severe). Scores are averaged to achieve a final score with a range of 0 to 4. Higher scores indicate greater frequency and severity of coercive controlling IPV.
Change in Child Anxiety Symptoms | Baseline, 19 weeks, 43 weeks and 70 weeks
  The Child Trauma Symptom Checklist will be used to assess child Anxiety symptoms. Each symptom item is rated according to its frequency of occurrence using a four point scale ranging from 0 ("never") to 3 ("often"). The Anxiety subscale score is converted to a t-score based on measure norms with scores ranging from 0 to 100. Higher scores indicate greater severity of anxiety symptoms.
Change in Child Depression Symptoms | Baseline, 19 weeks, 43 weeks and 70 weeks
  The Child Trauma Symptom Checklist will be used to assess child Depression symptoms. Each symptom item is rated according to its frequency of occurrence using a four point scale ranging from 0 ("never") to 3 ("often"). The depression subscale score is converted to a t-score based on measure norms with scores ranging from 0 to 100. Higher scores indicate greater severity of anxiety symptoms.
Change in Child Aggression Symptoms | Baseline, 19 weeks, 43 weeks and 70 weeks
  The Child Trauma Symptom Checklist will be used to assess child aggression symptoms. Each symptom item is rated according to its frequency of occurrence using a four point scale ranging from 0 ("never") to 3 ("often"). The Aggression subscale score is converted to a t-score based on measure norms with scores ranging from 0 to 100. Higher scores indicate greater severity of aggression symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Carla S Stover, PhD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale, New Haven, Connecticut
  - UCONN Health Center, West Hartford, Connecticut

IPD SHARING:
Plan to Share IPD: No